CLINICAL TRIAL: NCT07372989
Title: A Phase 1, Study of Nebulized Matrix - Allogeneic Human Amniotic Fluid (HAF) In Patients With Interstitial Lung Disease: AIRMID Trial
Brief Title: Nebulized Human Amniotic Fluid in Patients With Interstitial Lung Disease
Acronym: HAF ILD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Maule Stem Cell Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-MSCRI-001
Record Dates: First submitted 2026-01-14; First posted 2026-01-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lung Diseases, Interstitial
Keywords: Interstitial Lung Disease (ILD)
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: Participants will be placed into 2 Cohorts of 22 participants in each treatment arm:
  Cohort A: Doses 1.0 ml of Matrix 1×10^9 particles via mesh nebulizer
  Cohort B: Doses 1.5 ml of Matrix 1×10^12 particles via mesh nebulizer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): 1.0 mL of Matrix (Exosomes)
  Interventions: Biological: Matrix
- Cohort B (Experimental): 1.5 mL of Matrix (Exosomes)
  Interventions: Biological: Matrix

INTERVENTIONS:
Biological: Matrix — Allogeneic Human Amniotic Fluid (HAF) using Aerogen Solo (Ultra Nebulizer)

SUMMARY:
This is a Phase I, pilot clinical trial designed to evaluate the safety and exploratory efficacy of nebulized diluted amniotic fluid, Matrix (HAF-Matrix) in adults with interstitial lung disease (ILD). ILDs are progressive fibrotic disorders characterized by aberrant wound-healing responses, chronic inflammation, and dysregulated fibroblast activation, ultimately leading to impaired gas exchange and respiratory failure. Current treatments, such as antifibrotic agents (pirfenidone and nintedanib), slow disease progression but do not reverse existing fibrosis or restore lung function. This pilot study will generate critical safety and preliminary efficacy data to inform future larger-scale trials and optimize dosing strategies for nebulized HAF-based therapeutics in ILD.

DETAILED DESCRIPTION:
This pilot study will generate critical safety and preliminary efficacy data to inform future larger-scale trials and optimize dosing strategies for nebulized EV-based therapeutics in ILD.

Two-part seamless design:

Dose Escalation Approach with a 3+3 (Cohort A = 3, Cohort B = 3) Total of 6 Participants Design with Staggered Dosing:

1. Cohort Enrollment and Initial Dosing

• At each prespecified dose level, three (3) subjects will be enrolled and dosed.

The first subject in each cohort will be dosed initially, followed by the second and third subjects according to planned staggered intervals, ensuring careful monitoring of early safety signals.

Post 3x3 run-in phase, The Phase 1(open label) will begin:

* 2 Cohorts of 22 participants per cohort:
* Doses 1.0 ml and 1.5 ml of Matrix via mesh nebulizer:

Cohort A, n=22: 1×10^9 particles Cohort B, n=22: 1×10^12 particles (Dose range anchored to inhaled-EV clinical experience.)

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, a patient MUST:

* Provide written informed consent.
* Subjects age > 40 and < 90 years at the time of signing the Informed Consent Form.
* Have a clinical diagnosis of ILD prior to screening in accordance with the guidelines of the American Thoracic Society/European Respiratory Society.
* FVC ≥ 45% predicted and DLCO ≥30% (corrected for hemoglobin but not alveolar volume).
* Resting SpO₂ ≥ 92% on ≤ 3 L/min O₂.
* RVSP < 50 mmHg, as documented by Doppler echo or right heart catheterization.
* Female subjects must be surgically sterile or post-menopausal (>1 year).

Exclusion Criteria:

In order to participate in this study, a patient MUST NOT:

* CT and/or surgical lung biopsy results inconsistent with the diagnosis of IPF.
* Inability to perform any of the assessments required for endpoint analysis (report safety or tolerability concerns, perform PFTs or CT, undergo blood draws, read and respond to questionnaires.)
* Currently receiving (or received within four weeks of screening) any medication, treatment, or experimental agents for the treatment of ILD, except for patients receiving non-drug therapies will include oxygen saturation therapy (oxygen supplementation) and pulmonary rehabilitation.
* Active listing (or expected future listing) for transplant of any organ.
* Clinically important abnormal screening laboratory values, including but not limited to: hemoglobin <8 g/dl, white blood cell count <3000/mm3, platelets <80,000/mm3, INR > 1.5, aspartate transaminase, alanine transaminase, or alkaline phosphatase > 2 times upper limit of normal, total bilirubin > 1.5 mg/dl.
* Serious comorbid illness that, in the opinion of the investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study. Including, but not limited to: HIV, advanced liver or renal failure, class III/IV congestive heart failure, myocardial infarction, unstable angina, or cardiac revascularization within the last six months, or severe obstructive ventilatory defect.
* Any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study.
* Be an organ transplant recipient.
* Have a clinical history of malignancy within 2.5 years (i.e., patients with prior malignancy must be disease free for 2.5 years), except curatively treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma.
* Have a non-pulmonary condition that limits lifespan to < 1 year.
* Have a history of drug or alcohol abuse within the past 24 months.
* Be serum positive for HIV, hepatitis BsAg or Viremic hepatitis C.
* Be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial.
* Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods. Female patients must undergo a blood or urine pregnancy test at screening and within 36 hours prior to injection.
* Female subjects must have an FSH < 25.8 IU/L
* Subject with hypersensitivity to dimethyl sulfoxide (DMSO)
* Saturated oxygen (SpO2 of < 93% (room air [sea level] at rest). SpO2 of < 88% (room air [>5,000 feet above sea level (1524 meters) at rest).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From first dose through study completion (approximately 13 months)
  Outcome Measure Description:
  Incidence of treatment-emergent serious adverse events (TE-SAEs) in participants receiving nebulized Matrix (HAF) therapy.
  Unit of Measure:
  Number of participants with ≥1 TESAE

SECONDARY OUTCOMES:
Change in observed forced vital capacity (FVC) . | Baseline to 6 months.
  Change From Baseline in Forced Vital Capacity (FVC)
  Outcome Measure Description:
  Change from baseline in forced vital capacity (FVC) as assessed by pulmonary function testing.
  Unit of Measure:
  Liters (L) or percent predicted (%)

OTHER OUTCOMES:
Forced expiratory volume in 1 second (FEV1). | Baseline to 6 months
  Change From Baseline in Forced Expiratory Volume in 1 Second (FEV₁)
  Outcome Measure Description:
  Change from baseline in forced expiratory volume in 1 second (FEV₁) as assessed by pulmonary function testing.
  Unit of Measure:
  Liters (L) or percent predicted (%)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia S. Maule, M.D., Principal Investigator — Maule Stem Cell Research Institute
Locations (1):
- Maule Stem Cell Research Institute, Venice, Florida, United States

IPD SHARING:
Plan to Share IPD: No